CLINICAL TRIAL: NCT01313676
Title: A Clinical Outcomes Study to Compare the Effect of Fluticasone Furoate/Vilanterol Inhalation Powder 100/25mcg With Placebo on Survival in Subjects With Moderate Chronic Obstructive Pulmonary Disease (COPD) and a History of or at Increased Risk for Cardiovascular Disease
Brief Title: Study to Evaluate the Effect of Fluticasone Furoate/Vilanterol on Survival in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113782
Record Dates: First submitted 2011-02-03; First posted 2011-03-14 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Cardiovascular disease; Novel Dry Powder Inhaler; Survival
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- fluticasone furoate/vilanterol (Experimental): Combination of both products in one inhaler
  Interventions: Drug: fluticasone furoate/vilanterol
- fluticasone furoate (Experimental): comparator of individual component
  Interventions: Drug: fluticasone furoate
- vilanterol (Experimental): comparator of individual component
  Interventions: Drug: vilanterol
- placebo (Placebo Comparator): once daily via inhaler
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: fluticasone furoate/vilanterol — 100/25mcg given once daily via novel dry powder inhaler
  Arms: fluticasone furoate/vilanterol
Drug: fluticasone furoate — 100mcg given once daily via novel dry powder inhaler
  Arms: fluticasone furoate
Drug: vilanterol — 25mcg given once daily via novel dry powder inhaler
  Arms: vilanterol
Other: Placebo — placebo comparator once daily via novel dry powder inhaler
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if fluticasone furoate/vilanterol improves survival in patients with chronic obstructive pulmonary disease with a history of or increased risk of heart disease.

DETAILED DESCRIPTION:
Despite a potential link between the pathogenetic mechanisms involved in Chronic Obstructive Pulmonary Disease (COPD) and atherosclerotic cardiovascular disease, there are no currently approved therapies for patients with COPD that have clearly shown an additional beneficial effect in patients with cardiovascular comorbidities. The TOwards a Revolution in COPD Health (TORCH) study assessed the impact of the inhaled corticosteroid (ICS) fluticasone propionate (FP) in combination with the long-acting beta agonist (LABA), salmeterol (SAL), in reducing all-cause mortality. TORCH demonstrated a 17.5% reduction on all-cause mortality with salmeterol-fluticasone propionate combination (SFC) compared with placebo (HR=0.825, 95% CI (0.681, 1.002), p=0.052) in the entire COPD population with disease severity form moderate to very severe. A post hoc analysis of the data restricted to those subjects with an forced expiratory volume in 1 second (FEV1) >=50% predicted with an apparent history of cardiovascular co-morbidities (defined as use at baseline of beta-blockers, angiotensin converting enzyme inhibitors (ACEI)/angiotensin receptor blockers (ARB), HMG CoA reductase inhibitors (i.e. statins) or a prior MI recorded at baseline) demonstrated a 49% reduction in the risk of dying within 96 weeks for the comparison of SFC with placebo. These post hoc data suggest the possibility of an ICS/LABA combination product to be of substantial benefit in COPD subjects with less severe airflow obstruction yet with increased cardiovascular risk.

The mechanism by which SFC appears to be associated with a greater reduction in mortality in these less severe COPD subjects with concomitant cardiovascular comorbidities is speculative at present, but could potentially in part be related to a lessening of the degree of inflammation in the systemic circulation, potential plaque stabilization and/or amelioration of arterial stiffness.

ICS/LABA combinations that are currently available require twice daily administration. A once daily ICS/LABA combination has the potential to improve patient compliance and as a result, overall disease management.

The purpose of this study is to prospectively evaluate the effect of the once daily ICS/LABA combination Fluticasone Furoate (FF)/Vilanterol (VI) on survival in subjects with moderate COPD (>=50 and =<70 % predicted FEV1 ) and a history of, or at increased risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient.
* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Male or female. Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy. The decision to include or exclude women of childbearing potential may be made at the discretion of the investigator in accordance with local practice in relation to adequate contraception.
* Age: >=40 and <=80 years of age at Screening (Visit 1).
* Tobacco use: Subjects with a current or prior history of >=10 pack-years of cigarette smoking at screening (Visit 1). Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Airflow Obstruction:

Subjects with a measured post-albuterol/salbutamol forced expiratory volume in 1 second (FEV1)/(forced vital capacity)FVC ratio of <=0.70 at Screening (Visit 1).

Subjects with a measured post-albuterol/salbutamol FEV1 >=50 and <=70% of predicted normal values calculated using NHANES III reference equations [Hankinson, 1999; Hankinson, 2010] at Screening (Visit 1).

Post-bronchodilator spirometry will be performed approximately 15 minutes after the subject has self-administered 4 inhalations (i.e., total 400mcg) of albuterol/salbutamol via a metered dose inhaler (MDI )with a valved-holding chamber. The FEV1/FVC ratio and FEV1 percent predicted values will be calculated.

* Symptoms of COPD: Subjects must score 2 or higher on the modified Medical Research Council Dyspnea scale (Visit 1)
* Cardiovascular disease:

For patients >= 40 years of age: any one of the following:

Established (i.e. by clinical signs or imaging studies) coronary artery disease (CAD) Established (i.e. by clinical signs or imaging studies) peripheral vascular disease (PVD) Previous stroke Previous MI Diabetes mellitus with target organ disease OR

For patients >=60 years of age: any 2 of the following:

Being treated for hypercholesterolemia Being treated for hypertension Being treated for diabetes mellitus Being treated for peripheral vascular disease

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they also have a current diagnosis of COPD).
* alpha 1-antitrypsin deficiency: Subjects with known alpha-1 antitrypsin deficiency as the underlying cause of COPD.
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Lung resection or transplantation: Subjects with lung volume reduction surgery within the 12 months prior to Screening or having had a lung transplant.
* A moderate/severe COPD exacerbation that has not resolved at least 14 days prior to Visit 1 and at least 30 days following the last dose of oral corticosteroids (if applicable).
* Current severe heart failure (New York Heart Association class IV). Subjects will also be excluded if they have a known ejection fraction of <30% or if they have an implantable cardioverter defibrillator (ICD).
* Other diseases/abnormalities: Any life-threatening condition with life expectancy <3 years, other than vascular disease or COPD, that might prevent the subject from completing the study.
* End stage chronic renal disease: Subjects will be excluded if on renal replacement therapy (hemodialysis or peritoneal).
* Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroid) or components of the inhalation powder (e.g. lactose, magnesium stearate). In addition, patients with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e. <=12 hours per day) is not exclusionary.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study or the potential compliance to study procedures.
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.
* Additional medication: Use of the following medications within the following time intervals prior to Visit 1 or during the study (unless otherwise specified):

Medication No use within the following time intervals prior to Screening or thereafter at any time during the study (unless otherwise specified) Inhaled Long acting beta-agonists (LABA) 48 hours ICS/LABA combination products 48 hours Inhaled corticosteroids 48 hours Tiotropium 1 week Systemic, Oral, parenteral, intra-articular corticosteroids 30 days (oral and systemic corticosteroids may be used to treat COPD exacerbations during the study) Cytochrome P450 3A4 strong inhibitors including but not limited to antiretrovirals (protease inhibitors) (e.g.Indinavir, Nelfinavir, Ritonavir, Saquinavir); Imidazole and Triazole anti-fungals (e.g. Ketaconazole, Itraconazole); Clarithromycin, Telithromycin, Amiodarone, and Nefazodone 6 weeks Grapefruit is allowed up to Visit 1, then limited to no more than one glass of grapefruit juice (250 mL/ 8 ounces) or one grapefruit per day Any other investigational drug 30 days or 5 half lives whichever is longer.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16568 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1090):
- United States (372):
  - GSK Investigational Site, Andalusia, Alabama
  - GSK Investigational Site, Athens, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Ozark, Alabama
  - GSK Investigational Site, Pell City, Alabama
  - GSK Investigational Site, Tuscumbia, Alabama
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sierra Vista, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Gold River, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Lancaster, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Montclair, California
  - GSK Investigational Site, Monterey Park, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Pismo Beach, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Gabriel, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, San Marino, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Sepulveda, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Celebration, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Crystal River, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, DeBary, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fleming Island, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Leesburg, Florida
  - GSK Investigational Site, Lehigh Acres, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Gardens, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Summerfield, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Trinity, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Calhoun, Georgia
  - GSK Investigational Site, Canton, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Cumming, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Rincon, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Hayden Lake, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Quincy, Illinois
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Elwood, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Franklin, Indiana
  - GSK Investigational Site, Greenfield, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Olathe, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Hawesville, Kentucky
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Opelousas, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Biddeford, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Elkton, Maryland
  - GSK Investigational Site, Hagerstown, Maryland
  - GSK Investigational Site, Hollywood, Maryland
  - GSK Investigational Site, Lutherville, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Buckley, Michigan
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Rochester, Michigan
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Coon Rapids, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Freehold, New Jersey
  - GSK Investigational Site, Linden, New Jersey
  - GSK Investigational Site, Lodi, New Jersey
  - GSK Investigational Site, Margate City, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Salem, New Jersey
  - GSK Investigational Site, Verona, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Corning, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhattan, New York
  - GSK Investigational Site, Massapequa, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Knightdale, North Carolina
  - GSK Investigational Site, Lexington, North Carolina
  - GSK Investigational Site, Morganton, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Smithfield, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Chardon, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Marion, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Miamisburg, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Wooster, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Springfield, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Belle Vernon, Pennsylvania
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Clairton, Pennsylvania
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Harleysville, Pennsylvania
  - GSK Investigational Site, Jersey Shore, Pennsylvania
  - GSK Investigational Site, Langhorne, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Monroeville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Phoenixville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Scottdale, Pennsylvania
  - GSK Investigational Site, Scranton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Johnston, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Florence, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greenwood, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, Old Point Station, South Carolina
  - GSK Investigational Site, Pelzer, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Williamston, South Carolina
  - GSK Investigational Site, Dakota Dunes, South Dakota
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Fayetteville, Tennessee
  - GSK Investigational Site, Franklin, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Shelbyville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, Edinburg, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Frisco, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Huntsville, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Victoria, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Midvale, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Burien, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Bridgeport, West Virginia
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, West Allis, Wisconsin
- Argentina (40):
  - GSK Investigational Site, Adrogué, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Ciudad Autnónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Derqui, Pilar, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Olivos, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, San Isidro, Buenos Aires
  - GSK Investigational Site, San Juan Bautista, Buenos Aires
  - GSK Investigational Site, San Martín, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Vicente López, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, Paraná, Entre Ríos Province
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, Cipoletti, Rio Negro, Río Negro Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Coronel Suárez
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Formosa
  - GSK Investigational Site, Lanús
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Monte Grande
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Salta
  - GSK Investigational Site, San Juan Bautista
  - GSK Investigational Site, San Luis
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, San Salvador de Jujuy
  - GSK Investigational Site, Santa Fe
  - GSK Investigational Site, Santiago del Estero
- Australia (8):
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Redcliffe, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Glen Osmond
- Austria (11):
  - GSK Investigational Site, Feldbach
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Grieskirchen
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Spittal/Drau
  - GSK Investigational Site, Thalheim bei Wels
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wels
  - GSK Investigational Site, Zwettl Stadt
- Belarus (5):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Grodno
  - GSK Investigational Site, Homyel
  - GSK Investigational Site, Minsk
  - GSK Investigational Site, Vitebsk
- Belgium (5):
  - GSK Investigational Site, Diest
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Gilly
  - GSK Investigational Site, Mons
  - GSK Investigational Site, Namur
- Bosnia and Herzegovina (21):
  - GSK Investigational Site, Banja Luka
  - GSK Investigational Site, Bihać
  - GSK Investigational Site, Bijeljina
  - GSK Investigational Site, Brčko
  - GSK Investigational Site, Foča
  - GSK Investigational Site, Gračanica
  - GSK Investigational Site, Gradiška
  - GSK Investigational Site, Istocno Sarajevo
  - GSK Investigational Site, Konjic
  - GSK Investigational Site, Mostar
  - GSK Investigational Site, Novi Travnik
  - GSK Investigational Site, Pale
  - GSK Investigational Site, Sarajevo
  - GSK Investigational Site, Srebrenik
  - GSK Investigational Site, Teslić
  - GSK Investigational Site, Tešanj
  - GSK Investigational Site, Travnik
  - GSK Investigational Site, Trebinje
  - GSK Investigational Site, Tuzla
  - GSK Investigational Site, Višegrad
  - GSK Investigational Site, Zenica
- Bulgaria (19):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Kozloduy
  - GSK Investigational Site, Lovech
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Petrich
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Razgrad
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Troyan Municipality
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
  - GSK Investigational Site, Vidin
- Canada (20):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kamloops, British Columbia
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, West Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Bolton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Orléans, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
- Chile (3):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (34):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Hohhot, Hainan
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Baotou, Inner Mongolia
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Baotou
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Bengbu
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangxi
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Huai'an
  - GSK Investigational Site, Jiangyin
  - GSK Investigational Site, Luzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuxi
- Colombia (5):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Medellín
  - GSK Investigational Site, Zipaquirá
- Croatia (25):
  - GSK Investigational Site, Čakovec
  - GSK Investigational Site, Draganići
  - GSK Investigational Site, Hrašće Turopoljsko
  - GSK Investigational Site, Hreljin
  - GSK Investigational Site, Ivankovo
  - GSK Investigational Site, Karlovac
  - GSK Investigational Site, Klenovnik
  - GSK Investigational Site, Krapina
  - GSK Investigational Site, Kutina
  - GSK Investigational Site, Novi Marof
  - GSK Investigational Site, Osijek
  - GSK Investigational Site, Retkovci
  - GSK Investigational Site, Rijeka
  - GSK Investigational Site, Samobor
  - GSK Investigational Site, Senj
  - GSK Investigational Site, Sisak
  - GSK Investigational Site, Split
  - GSK Investigational Site, Strmec
  - GSK Investigational Site, Stubičke Toplice
  - GSK Investigational Site, Sukosan
  - GSK Investigational Site, Šibenik
  - GSK Investigational Site, Varaždin
  - GSK Investigational Site, Zabok
  - GSK Investigational Site, Zadar
  - GSK Investigational Site, Zagreb
- Czechia (28):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Beroun
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Hlučín
  - GSK Investigational Site, Holešov
  - GSK Investigational Site, Jaroměř
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kolín
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Kroměříž
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Mělník
  - GSK Investigational Site, Moravský Krumlov
  - GSK Investigational Site, Neratovice
  - GSK Investigational Site, Nový Jičín
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Ostrava - Belsky Les
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Rudná
  - GSK Investigational Site, Strakonice
  - GSK Investigational Site, Svitavy
  - GSK Investigational Site, Třemošná
  - GSK Investigational Site, Usti Nad Labem - Klise
  - GSK Investigational Site, Žatec
- France (5):
  - GSK Investigational Site, Férolles-Attilly
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tarbes
  - GSK Investigational Site, Toulouse
- Georgia (5):
  - GSK Investigational Site, Batumi
  - GSK Investigational Site, Gurjaani
  - GSK Investigational Site, Kutaisi
  - GSK Investigational Site, Kvemo Kartli
  - GSK Investigational Site, Tbilisi
- Germany (58):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Ettlingen, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Feldkirchen, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Höchstadt an der Aisch, Bavaria
  - GSK Investigational Site, Landsberg am Lech, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Vilshofen, Bavaria
  - GSK Investigational Site, Weißenhorn, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Bensheim, Hesse
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Papenburg, Lower Saxony
  - GSK Investigational Site, Stuhr, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Hagen, North Rhine-Westphalia
  - GSK Investigational Site, Harsewinkel, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Föhren, Rhineland-Palatinate
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Neuwied, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Görlitz, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Riesa, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Hungary (18):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Komárom
  - GSK Investigational Site, Komló
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Nagykanizsa
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Sopron
  - GSK Investigational Site, Szigetszentmiklós
  - GSK Investigational Site, Szikszó
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Tatabánya
  - GSK Investigational Site, Vásárosnamény
  - GSK Investigational Site, Zalaegerszeg
- India (18):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Alappuzha
  - GSK Investigational Site, Angamaly
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Guntur
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Mysore
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trisshur
  - GSK Investigational Site, Trivandrum
  - GSK Investigational Site, Varanasi
  - GSK Investigational Site, Vijayawada
- Indonesia (19):
  - GSK Investigational Site, Banda Aceh
  - GSK Investigational Site, Banjarmasin
  - GSK Investigational Site, Bukittinggi
  - GSK Investigational Site, Denpasar
  - GSK Investigational Site, Depok Timur
  - GSK Investigational Site, Jakarta
  - GSK Investigational Site, Lampung Selatan
  - GSK Investigational Site, Makassar
  - GSK Investigational Site, Malang
  - GSK Investigational Site, Medan
  - GSK Investigational Site, Padang
  - GSK Investigational Site, Palembang
  - GSK Investigational Site, Pekanbaru
  - GSK Investigational Site, Pontianak
  - GSK Investigational Site, Pringsewu
  - GSK Investigational Site, Semarang
  - GSK Investigational Site, Surabaya
  - GSK Investigational Site, Surakarta
  - GSK Investigational Site, Yogyakarta
- Israel (11):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Hadera
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Tel Litwinsky
- GSK Investigational Site, Pordenone, Friuli Venezia Giulia, Italy
- Japan (14):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kodaira
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Tokyo
- Latvia (14):
  - GSK Investigational Site, Balvi
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Jelgava
  - GSK Investigational Site, Jēkabpils
  - GSK Investigational Site, Jūrmala
  - GSK Investigational Site, Krāslava
  - GSK Investigational Site, Kuldīga
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Ogre
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Talsi
  - GSK Investigational Site, Tukums
  - GSK Investigational Site, Valmiera
  - GSK Investigational Site, Ventspils
- Malaysia (8):
  - GSK Investigational Site, Johor Bahru
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Pilah
  - GSK Investigational Site, Kuala Selangor
  - GSK Investigational Site, Kuching
  - GSK Investigational Site, Sibu
  - GSK Investigational Site, Sungai Petani, Kedah
  - GSK Investigational Site, Taiping Perak
- Mexico (16):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Hermosillo, Sonora
  - GSK Investigational Site, Cuautitlán Izcalli, State of Mexico
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Hidalgo
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, México DF
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, San Luis Potosí City
- Netherlands (5):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Ede Gld
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Zutphen
- North Macedonia (8):
  - GSK Investigational Site, Bitola
  - GSK Investigational Site, Gostivar
  - GSK Investigational Site, Ohrid
  - GSK Investigational Site, Prilep
  - GSK Investigational Site, Shtip
  - GSK Investigational Site, Skopje
  - GSK Investigational Site, Strumica
  - GSK Investigational Site, Veles
- Philippines (16):
  - GSK Investigational Site, Alabang, Muntinlupa City
  - GSK Investigational Site, Caloocan
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Los Baños
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marilao, Bulacan
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Fernando, Pampanga
- Poland (59):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Bieńkówka
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chełmża
  - GSK Investigational Site, Chodzież
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Choszczno
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Dąbrowa Górnicza
  - GSK Investigational Site, Działdowo
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Gorzów Wielkopolski
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Izabelin
  - GSK Investigational Site, Iława
  - GSK Investigational Site, Jelenia Góra
  - GSK Investigational Site, Karpacz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Krotoszyn
  - GSK Investigational Site, Ksawerów
  - GSK Investigational Site, Kutno
  - GSK Investigational Site, Libiąż
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Ostrow Wilekopolski
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Oława
  - GSK Investigational Site, Piaseczno
  - GSK Investigational Site, Piła
  - GSK Investigational Site, Police
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Płock
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Rudka
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Skarżysko-Kamienna
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Świdnik
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Tczew
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wodzisław Śląski
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Włocławek
  - GSK Investigational Site, Włoszczowa
  - GSK Investigational Site, Zabrze
  - GSK Investigational Site, Zgierz
  - GSK Investigational Site, Łęczyca
- Romania (17):
  - GSK Investigational Site, Arad
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bragadiru
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Campulung Muscel
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Târgu Mureş
  - GSK Investigational Site, Timișoara
- Russia (34):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kaliningrad
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kirov
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Pskov
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Sestroretsk
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, St.Рetersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Vsevolzhsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Serbia (7):
  - GSK Investigational Site, Belgrade
  - GSK Investigational Site, Čačak
  - GSK Investigational Site, Kamenitz
  - GSK Investigational Site, Kragujevac
  - GSK Investigational Site, Niš
  - GSK Investigational Site, Sombor
  - GSK Investigational Site, Valjevo
- Slovakia (9):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Kráľovský Chlmec
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Spišská Nová Ves
  - GSK Investigational Site, Štúrovo
  - GSK Investigational Site, Trnava
  - GSK Investigational Site, Vráble
- South Africa (28):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, Morningside, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Thaba Tshwane, Gauteng
  - GSK Investigational Site, Dundee, KwaZulu-Natal
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, CapeTown
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Korsten
  - GSK Investigational Site, Lynnwood Ridge
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Potchefstroom
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Roodepoort
  - GSK Investigational Site, Rooihuiskraal
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Thabazimbi
  - GSK Investigational Site, Tygerberg
  - GSK Investigational Site, Voorspoed
- South Korea (19):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Bucheon-Si, Gyeonggi-Do
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Cheonan
  - GSK Investigational Site, Chonju-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Goyang-si
  - GSK Investigational Site, Guri-si
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon
  - GSK Investigational Site, Seongnam
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Gyeonggi-do
  - GSK Investigational Site, Uijeongbu, Gyeonggi-do
  - GSK Investigational Site, Ulsan
  - GSK Investigational Site, Wonju-si, Kanwon-do
- Spain (22):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benidorm
  - GSK Investigational Site, Canet de Mar - Barcelona
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Illescas-Toledo
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, Sant Boi de Llobregat
  - GSK Investigational Site, Santa Coloma de Gramenet
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Torrelavega
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic (Barcelona)
- Taiwan (10):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Chiayi City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Kaohsiung Hsien
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, Linkou District
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Yung Kang City
- Thailand (9):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Chiangrai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Mae Rim, Chiang Mai
  - GSK Investigational Site, Muang
  - GSK Investigational Site, Nakhon Ratchasima
  - GSK Investigational Site, Phitsanulok
  - GSK Investigational Site, Songkhla
- Turkey (Türkiye) (6):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Bursa
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Kocaeli
  - GSK Investigational Site, Konya
  - GSK Investigational Site, Samsun
- Ukraine (28):
  - GSK Investigational Site, Alupka
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Chernihiv
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kherson
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kryvyi Rig
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lutsk
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Sympheropol
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Yalta
  - GSK Investigational Site, Zaporizhia
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zaporizhzhya
  - GSK Investigational Site, Zhytomyr
- United Kingdom (24):
  - GSK Investigational Site, Bedford, Bedfordshire
  - GSK Investigational Site, Peterborough, Cambridgeshire
  - GSK Investigational Site, Soham, Cambridgeshire
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Waterloo, Liverpool, Merseyside
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Bury St Edmunds, Suffolk
  - GSK Investigational Site, Bexhill-on-Sea
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Derby
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Milton Keynes
  - GSK Investigational Site, Reading
  - GSK Investigational Site, Sidcup, Kent
  - GSK Investigational Site, Tyne and Wear
- Vietnam (4):
  - GSK Investigational Site, Can Tho
  - GSK Investigational Site, Hà Nội
  - GSK Investigational Site, Ho Chi Minh City
  - GSK Investigational Site, Huế

REFERENCES:
- [Derived] Verstraete K, Gyselinck I, Huts H, Das N, Topalovic M, De Vos M, Janssens W. Estimating individual treatment effects on COPD exacerbations by causal machine learning on randomised controlled trials. Thorax. 2023 Oct;78(10):983-989. doi: 10.1136/thorax-2022-219382. Epub 2023 Apr 3. PMID 37012070
- [Derived] Horne BD, Hegewald MJ, Crim C, Rea S, Bair TL, Blagev DP. The Summit Score Stratifies Mortality and Morbidity in Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 Jul 20;15:1741-1750. doi: 10.2147/COPD.S254437. eCollection 2020. PMID 32764918
- [Derived] Wise RA, Anderson JA, Amarenco P, Cowans NJ, Crim C, Denvir MA, Gomez CR, Jones MP, Morris A, Niewoehner D, Yates JC. Adjudication of cardiovascular events in patients with chronic obstructive pulmonary disease: SUMMIT trial. Clin Trials. 2020 Aug;17(4):430-436. doi: 10.1177/1740774520920897. Epub 2020 May 22. PMID 32441114
- [Derived] Celli BR, Anderson JA, Brook R, Calverley P, Cowans NJ, Crim C, Dixon I, Kim V, Martinez FJ, Morris A, Newby DE, Yates J, Vestbo J. Serum biomarkers and outcomes in patients with moderate COPD: a substudy of the randomised SUMMIT trial. BMJ Open Respir Res. 2019 May 4;6(1):e000431. doi: 10.1136/bmjresp-2019-000431. eCollection 2019. PMID 31258919
- [Derived] Fawzy A, Anderson JA, Cowans NJ, Crim C, Wise R, Yates JC, Hansel NN. Association of platelet count with all-cause mortality and risk of cardiovascular and respiratory morbidity in stable COPD. Respir Res. 2019 May 8;20(1):86. doi: 10.1186/s12931-019-1059-1. PMID 31068182
- [Derived] Vestbo J, Dransfield M, Anderson JA, Brook RD, Calverley PMA, Celli BR, Cowans NJ, Crim C, Martinez F, Newby DE, Yates J, Lange P. Impact of pre-enrolment medication use on clinical outcomes in SUMMIT. ERJ Open Res. 2019 Feb 25;5(1):00203-2018. doi: 10.1183/23120541.00203-2018. eCollection 2019 Feb. PMID 30815468
- [Derived] Adamson PD, Anderson JA, Brook RD, Calverley PMA, Celli BR, Cowans NJ, Crim C, Dixon IJ, Martinez FJ, Newby DE, Vestbo J, Yates JC, Mills NL. Cardiac Troponin I and Cardiovascular Risk in Patients With Chronic Obstructive Pulmonary Disease. J Am Coll Cardiol. 2018 Sep 4;72(10):1126-1137. doi: 10.1016/j.jacc.2018.06.051. PMID 30165984
- [Derived] Kunisaki KM, Dransfield MT, Anderson JA, Brook RD, Calverley PMA, Celli BR, Crim C, Hartley BF, Martinez FJ, Newby DE, Pragman AA, Vestbo J, Yates JC, Niewoehner DE; SUMMIT Investigators. Exacerbations of Chronic Obstructive Pulmonary Disease and Cardiac Events. A Post Hoc Cohort Analysis from the SUMMIT Randomized Clinical Trial. Am J Respir Crit Care Med. 2018 Jul 1;198(1):51-57. doi: 10.1164/rccm.201711-2239OC. PMID 29442524
- [Derived] Celli B, Anderson JA, Brook R, Calverley P, Crim C, Holmes AP, Martinez FJ, Newby DE, Yates J, Vestbo J; SUMMIT Investigators. Long-Acting beta-Agonist/Inhaled Corticosteroid in Patients with Chronic Obstructive Pulmonary Disease with Cardiovascular Disease or Risk: A Factorial Analysis of the SUMMIT Clinical Trial. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1641-1644. doi: 10.1164/rccm.201710-2052LE. No abstract available. PMID 29412688
- [Derived] Dransfield MT, McAllister DA, Anderson JA, Brook RD, Calverley PMA, Celli BR, Crim C, Gallot N, Martinez FJ, Scanlon PD, Yates J, Vestbo J, Newby DE; SUMMIT Investigators. beta-Blocker Therapy and Clinical Outcomes in Patients with Moderate Chronic Obstructive Pulmonary Disease and Heightened Cardiovascular Risk. An Observational Substudy of SUMMIT. Ann Am Thorac Soc. 2018 May;15(5):608-614. doi: 10.1513/AnnalsATS.201708-626OC. PMID 29406772
- [Derived] Bhatt SP, Anderson JA, Brook RD, Calverley PMA, Celli BR, Cowans NJ, Crim C, Martinez FJ, Newby DE, Vestbo J, Yates JC, Dransfield MT. Cigarette smoking and response to inhaled corticosteroids in COPD. Eur Respir J. 2018 Jan 18;51(1):1701393. doi: 10.1183/13993003.01393-2017. Print 2018 Jan. No abstract available. PMID 29348179
- [Derived] Crim C, Calverley PMA, Anderson JA, Holmes AP, Kilbride S, Martinez FJ, Brook RD, Newby DE, Yates JC, Celli BR, Vestbo J; SUMMIT investigators. Pneumonia risk with inhaled fluticasone furoate and vilanterol in COPD patients with moderate airflow limitation: The SUMMIT trial. Respir Med. 2017 Oct;131:27-34. doi: 10.1016/j.rmed.2017.07.060. Epub 2017 Aug 1. PMID 28947039
- [Derived] Calverley PMA, Anderson JA, Brook RD, Crim C, Gallot N, Kilbride S, Martinez FJ, Yates J, Newby DE, Vestbo J, Wise R, Celli BR; SUMMIT (Study to Understand Mortality and Morbidity) Investigators. Fluticasone Furoate, Vilanterol, and Lung Function Decline in Patients with Moderate Chronic Obstructive Pulmonary Disease and Heightened Cardiovascular Risk. Am J Respir Crit Care Med. 2018 Jan 1;197(1):47-55. doi: 10.1164/rccm.201610-2086OC. PMID 28737971
- [Derived] Brook RD, Anderson JA, Calverley PM, Celli BR, Crim C, Denvir MA, Magder S, Martinez FJ, Rajagopalan S, Vestbo J, Yates J, Newby DE; SUMMIT Investigators. Cardiovascular outcomes with an inhaled beta2-agonist/corticosteroid in patients with COPD at high cardiovascular risk. Heart. 2017 Oct;103(19):1536-1542. doi: 10.1136/heartjnl-2016-310897. Epub 2017 Apr 17. PMID 28416587
- [Derived] Martinez FJ, Vestbo J, Anderson JA, Brook RD, Celli BR, Cowans NJ, Crim C, Dransfield M, Kilbride S, Yates J, Newby DE, Niewoehner D, Calverley PM; SUMMIT Investigators. Effect of Fluticasone Furoate and Vilanterol on Exacerbations of Chronic Obstructive Pulmonary Disease in Patients with Moderate Airflow Obstruction. Am J Respir Crit Care Med. 2017 Apr 1;195(7):881-888. doi: 10.1164/rccm.201607-1421OC. PMID 27767328
- [Derived] Vestbo J, Anderson JA, Brook RD, Calverley PM, Celli BR, Crim C, Martinez F, Yates J, Newby DE; SUMMIT Investigators. Fluticasone furoate and vilanterol and survival in chronic obstructive pulmonary disease with heightened cardiovascular risk (SUMMIT): a double-blind randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1817-26. doi: 10.1016/S0140-6736(16)30069-1. Epub 2016 Apr 28. PMID 27203508
- [Derived] Vestbo J, Anderson J, Brook RD, Calverley PM, Celli BR, Crim C, Haumann B, Martinez FJ, Yates J, Newby DE. The Study to Understand Mortality and Morbidity in COPD (SUMMIT) study protocol. Eur Respir J. 2013 May;41(5):1017-22. doi: 10.1183/09031936.00087312. Epub 2012 Sep 27. PMID 23018908
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1373 sites. The study employed an event-driven design and was to conclude when approximately 1000 reports of a primary outcome event of death were received. The study consisted of a 4-10 day run-in period, variable treatment period until the required number of events was achieved, and 1 week follow-up period.
Pre-assignment Details: A total of 23,835 participants were screened, of whom 16,590 were randomized. Of the 16,590 participants randomized, 16,568 participants received a single dose of investigational product (IP) and were assigned to a treatment and included in the Safety Population.
Groups:
- Placebo: Participants received placebo once daily (OD) in the morning from the dry powder inhaler (DPI) until the required number of events (death) was achieved. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- Fluticasone Furoate 100 µg: Participants received Fluticasone Furoate (FF) 100 microgram (µg) inhalation powder OD in the morning from the DPI until the required number of events (death) was achieved. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- Vilanterol 25 µg: Participants received Vilanterol (VI) 25 µg inhalation powder OD in the morning from the DPI until the required number of events (death) was achieved. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- Fluticasone Furoate/Vilanterol 100/25 µg: Participants received FF/VI 100/25 µg inhalation powder OD in the morning from the DPI until the required number of events (death) was achieved. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg
Started | 4131 | 4157 | 4140 | 4140
Completed | 2881 | 3044 | 3052 | 3146
Not Completed | 1250 | 1113 | 1088 | 994
Not completed — Adverse Event | 395 | 365 | 372 | 333
Not completed — Lack of Efficacy | 98 | 90 | 65 | 46
Not completed — Protocol Violation | 37 | 44 | 46 | 44
Not completed — Met Protocol-Defined Stopping Critera | 3 | 4 | 2 | 11
Not completed — Study Closed/terminated | 7 | 6 | 9 | 9
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 53 | 64 | 62 | 48
Not completed — Decision by Participant or Proxy | 643 | 527 | 515 | 492
Not completed — Sponsor Terminated Study Treatment | 1 | 1 | 0 | 1
Not completed — Investigator Site Closed | 12 | 11 | 15 | 10
Not completed — Missing | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg | Total
Number analyzed (Participants) | 4131 | 4157 | 4140 | 4140 | 16568
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (7.90) | 65.0 (8.02) | 65.2 (7.68) | 65.3 (7.97) | 65.2 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1050 | 1098 | 1071 | 1019 | 4238
  Male | 3081 | 3059 | 3069 | 3121 | 12330
Race/Ethnicity, Customized [Number; unit: Participants]
  African American /African Heritage | 61 | 62 | 68 | 69 | 260
  American Indian or Alaskan Native | 9 | 5 | 4 | 9 | 27
  Asian - Central /South Asian Heritage | 64 | 55 | 62 | 57 | 238
  Asian - East Asian Heritage | 192 | 193 | 195 | 192 | 772
  Asian - Japanese Heritage | 34 | 36 | 37 | 37 | 144
  Asian - Mixed Race | 1 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 389 | 399 | 386 | 394 | 1568
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 2 | 5
  White - Arabic/North African Heritage | 14 | 13 | 7 | 12 | 46
  White - Mixed Race | 0 | 0 | 0 | 1 | 1
  White - White/Caucasian /European Heritage | 3334 | 3367 | 3353 | 3337 | 13391
  Mixed Race | 32 | 25 | 28 | 30 | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death (Both on and Off Treatment) Due to Any Cause, Time up to or on the Pre-determined Common End Date
Description: Death from any cause: which occurred from the day of starting IP until the Commone End Date (CED). Common End Date (CED) is the study end date that was pre determined where approximately 1000 deaths would have occurred in the Intent-toTreat Efficacy (ITT-E) Population. Only deaths which occurred on or before the CED were used for the primary analysis. Those who had not died by CED, but who were known to be alive on or after the CED, were censored at the CED. Cox Proportional Hazards (PH) Model was adjusted for age, and gender, including all 4 arms. A hazard ratio of less than 1 indicates a lower death rate versus placebo or other arm. ITT-E Population consisted of all participants in the Safety Population (i.e. randomized to IP and who received at least one dose of IP), with the exception of those recruited at sites that were closed.
Time Frame: From the date of randomization until date of death due to any cause (average of 2 study years)
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg
Number analyzed (Participants) | 4111 | 4135 | 4118 | 4121
Participants
  Dead | 275 | 251 | 265 | 246
  Alive | 3832 | 3884 | 3853 | 3874
  Unknown | 4 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.137, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.739 to 1.042]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 12.2, 95% CI 2-sided [-4.2 to 26.1] — Confidence Interval (95%) and Estimated Value is presented for the percent reduction in risk of death at any time up to or on the CED, calculated as (1-hazard ratio)*100
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 100 µg; Test type: Superiority or Other; p = 0.284, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.911, 95% CI 2-sided [0.767 to 1.081]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate 100 µg; Test type: Superiority or Other; Percent reduction in risk of death = 8.9, 95% CI 2-sided [-8.1 to 23.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Vilanterol 25 µg; Test type: Superiority or Other; p = 0.655, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.962, 95% CI 2-sided [0.813 to 1.139]
Statistical Analysis 6: Comparison: Placebo vs Vilanterol 25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 3.8, 95% CI 2-sided [-13.9 to 18.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Fluticasone Furoate 100 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.681, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.964, 95% CI 2-sided [0.808 to 1.149]
Statistical Analysis 8: Comparison: Fluticasone Furoate 100 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 3.6, 95% CI 2-sided [-14.9 to 19.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Vilanterol 25 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.299, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.912, 95% CI 2-sided [0.767 to 1.085]
Statistical Analysis 10: Comparison: Vilanterol 25 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 8.8, 95% CI 2-sided [-8.5 to 23.3] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Decline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The effect of treatment on decline of post bronchodilator FEV1 recorded during the treatment period was analyzed using a particular form of a mixed effect model - a random coefficients model. FEV1 was fitted as the response variable with treatment group, age, gender, baseline FEV1 and time on treatment as fixed effects. Time on treatment was treated as a continuous variable. This model allowed for an initial increase in FEV1, but then tested the difference in slopes from the first post-baseline measurement which was at 3 months. A negative slope indicates a decline. A positive treatment difference indicates a slower rate of decline vs Placebo or Component. Only participants with at least one on-treatment post-bronchodilator FEV1 measurement were analyzed.
Time Frame: From start date of IP until IP stop date + 1 (assessed up to 4 years)
Population: ITT-E Population
Measure: Least Squares Mean (Standard Error); unit: milliliter/year
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg
Number analyzed (Participants) | 3800 | 3879 | 3866 | 3912
milliliter/year | -46 (2.5) | -38 (2.4) | -47 (2.4) | -38 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = 8, 95% CI 2-sided [1 to 15], Standard Error of Mean 3.4
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 100 µg; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 8, 95% CI 2-sided [1 to 14], Standard Error of Mean 3.5
Statistical Analysis 3: Comparison: Placebo vs Vilanterol 25 µg; Test type: Superiority or Other; p = 0.654, Mixed Models Analysis; Mean Difference (Final Values) = -2, 95% CI 2-sided [-8 to 5], Standard Error of Mean 3.4
Statistical Analysis 4: Comparison: Fluticasone Furoate 100 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.913, Mixed Models Analysis; Mean Difference (Final Values) = 0, 95% CI 2-sided [-6 to 7], Standard Error of Mean 3.4
Statistical Analysis 5: Comparison: Vilanterol 25 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 10, 95% CI 2-sided [3 to 16], Standard Error of Mean 3.4

3. Secondary Outcome: Number of Participants With First On-treatment Cardiovascular (CV) Composite Events Occured on or Before Common End Date
Description: On-treatment CV composite event is comprised of the first event that is adjudicated as on-treatment CV death, myocardial infarction, stroke, unstable angina, or transient ischemic attack experienced by a participant. The events that occurred no more than 7 days after the participants last dose of IP are considered as on-treatment adverse events. Common end date is the study end date where approximately 1000 deaths would have occurred in the ITT-E Population. Cox PH Model was used to assess time to first on-treatment CV composite event. Cox PH Model was adjusted for age, gender and indicators of ischemic and vascular disease, including all four treatment arms. A hazard ratio less than 1 indicates a lower risk of a first CV event rate versus placebo or any arm.
Time Frame: From the start of IP to first on treatment CV event till 7 days after the last dose of IP (average of 2 study years)
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg
Number analyzed (Participants) | 4111 | 4135 | 4118 | 4121
Participants
  Had CV composite event | 173 | 161 | 180 | 174
  No CV composite event | 3938 | 3974 | 3938 | 3947
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.475, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.926, 95% CI 2-sided [0.750 to 1.143]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; Percent reduction in risk of CV event = 7.4, 95% CI 2-sided [-14.3 to 25.0] — Confidence Interval and Estimated Value is presented for the percent reduction in risk of death at any time up to or on the CED, calculated as (1-hazard ratio)*100
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 100 µg; Test type: Superiority or Other; p = 0.317, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.896, 95% CI 2-sided [0.723 to 1.111]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate 100 µg; Test type: Superiority or Other; Percent reduction in risk of CV event = 10.4, 95% CI 2-sided [-11.1 to 27.7] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Vilanterol 25 µg; Test type: Superiority or Other; p = 0.908, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.988, 95% CI 2-sided [0.802 to 1.217]
Statistical Analysis 6: Comparison: Placebo vs Vilanterol 25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 1.2, 95% CI 2-sided [-21.7 to 19.8] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Fluticasone Furoate 100 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.763, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.033, 95% CI 2-sided [0.834 to 1.281]
Statistical Analysis 8: Comparison: Fluticasone Furoate 100 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; Percent reduction in risk of death = -3.3, 95% CI 2-sided [-28.1 to 16.6] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Vilanterol 25 µg vs Fluticasone Furoate/Vilanterol 100/25 µg; Test type: Superiority or Other; p = 0.545, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.938, 95% CI 2-sided [0.761 to 1.155]
Statistical Analysis 10: Comparison: Vilanterol 25 µg; Test type: Superiority or Other; Percent reduction in risk of death = 6.2, 95% CI 2-sided [-15.5 to 23.9] — [estimate comment as in outcome 3, analysis 2]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of IP until IP discontinuation + 1 day (average of 2 study years).
Description: On-treatment SAEs and non-serious AEs are reported for safety population, comprised of all participants randomized to treatment who received at least one dose IP.
Arm/Group | Placebo | Fluticasone Furoate 100 µg | Vilanterol 25 µg | Fluticasone Furoate/Vilanterol 100/25 µg
Serious Adverse Events (participants affected / at risk) | 918/4131 | 929/4157 | 972/4140 | 961/4140
Other Adverse Events (participants affected / at risk) | 1862/4131 | 1941/4157 | 1827/4140 | 1761/4140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4131) | Fluticasone Furoate 100 µg (N=4157) | Vilanterol 25 µg (N=4140) | Fluticasone Furoate/Vilanterol 100/25 µg (N=4140)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 3 | 5
Bone marrow oedema (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 3 | 6 | 5
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 23 | 20 | 21 | 28
Adams-Stokes syndrome (Cardiac disorders) | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 22 | 19 | 20 | 12
Angina unstable (Cardiac disorders) | 23 | 22 | 16 | 23
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 3
Arrhythmia (Cardiac disorders) | 1 | 4 | 3 | 6
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 1 | 1 | 3
Atrial fibrillation (Cardiac disorders) | 31 | 22 | 30 | 32
Atrial flutter (Cardiac disorders) | 6 | 3 | 3 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 2 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 3 | 2 | 3 | 3
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 2 | 3 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 3 | 1 | 1 | 3
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 9 | 9 | 11 | 4
Cardiac failure (Cardiac disorders) | 28 | 17 | 19 | 28
Cardiac failure acute (Cardiac disorders) | 7 | 3 | 3 | 7
Cardiac failure chronic (Cardiac disorders) | 5 | 7 | 4 | 7
Cardiac failure congestive (Cardiac disorders) | 26 | 26 | 21 | 30
Cardiac perforation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 11 | 9 | 11 | 5
Cardiogenic shock (Cardiac disorders) | 2 | 1 | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 2 | 4
Cardiopulmonary failure (Cardiac disorders) | 1 | 3 | 4 | 4
Cardiovascular disorder (Cardiac disorders) | 1 | 2 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 2 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 2 | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 2 | 0 | 2
Coronary artery disease (Cardiac disorders) | 22 | 14 | 25 | 24
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 3 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 2 | 1 | 2
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 4 | 3 | 4 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 3 | 2 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0 | 0 | 2
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 24 | 32 | 26 | 24
Myocardial ischaemia (Cardiac disorders) | 7 | 8 | 5 | 7
Myocardial necrosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 0
Rheumatic heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Sinoatrial block (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 3 | 2 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 3 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricle rupture (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 3 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 3 | 2 | 3
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Sturge-Weber syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 4 | 1 | 3
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1 | 1 | 0
Addison's disease (Endocrine disorders) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 3 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Primary hyperaldosteronism (Endocrine disorders) | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 5 | 8 | 6
Cataract cortical (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 1
Iridodonesis (Eye disorders) | 0 | 0 | 1 | 0
Lens dislocation (Eye disorders) | 1 | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 0
Ocular ischaemic syndrome (Eye disorders) | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 2 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1 | 0 | 0
Vitreous prolapse (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 5 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 1 | 6
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 4 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 5 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 4 | 4 | 4
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 5 | 2
Ileus paralytic (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 8 | 4 | 4 | 8
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 3 | 4
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 1 | 2 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 4 | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 4 | 7 | 2 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 2 | 2 | 3 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritoneal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 5 | 1 | 2
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 1 | 1
Cardiac death (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 3
Chest pain (General disorders) | 16 | 10 | 8 | 16
Cyst (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 6 | 7 | 5 | 7
Device defective (General disorders) | 0 | 0 | 0 | 1
Device deployment issue (General disorders) | 0 | 0 | 1 | 0
Device dislocation (General disorders) | 0 | 0 | 0 | 1
Device electrical finding (General disorders) | 0 | 1 | 0 | 0
Device failure (General disorders) | 1 | 0 | 0 | 0
Device issue (General disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 2 | 0 | 1 | 0
Device occlusion (General disorders) | 1 | 2 | 1 | 1
Electrocution (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 2 | 0 | 3 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Ischaemic ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Medical device complication (General disorders) | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 2 | 3 | 2 | 6
Non-cardiac chest pain (General disorders) | 4 | 5 | 10 | 3
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 1
Sudden cardiac death (General disorders) | 3 | 7 | 6 | 1
Sudden death (General disorders) | 20 | 14 | 17 | 20
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 0 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 7 | 4 | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 3 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 5 | 3 | 4 | 8
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 2 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 0
Acute hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 1 | 1 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 12 | 9 | 6 | 6
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 3 | 8 | 7 | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 5 | 10 | 0 | 6
Cholangitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 2 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 3 | 1 | 1
Diverticulitis (Infections and infestations) | 4 | 2 | 3 | 3
Embolic pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Emphysematous cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 3
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 3 | 3 | 1 | 2
Gastroenteritis (Infections and infestations) | 6 | 2 | 3 | 2
Gastroenteritis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Graft infection (Infections and infestations) | 0 | 0 | 1 | 1
Groin abscess (Infections and infestations) | 1 | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 3 | 2
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disea (Infections and infestations) | 4 | 6 | 3 | 6
Influenza (Infections and infestations) | 2 | 1 | 0 | 4
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 1
Lobar pneumonia (Infections and infestations) | 8 | 8 | 5 | 9
Lower respiratory tract infection (Infections and infestations) | 2 | 4 | 0 | 2
Lung abscess (Infections and infestations) | 0 | 2 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 1 | 0 | 0
Lymph node abscess (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 1 | 0 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 2 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 4 | 1 | 3
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 2 | 4 | 3
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 113 | 121 | 90 | 123
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 1 | 0 | 1
Pneumonia moraxella (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 1 — s
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 3 | 1 | 0 | 3
Purulent discharge (Infections and infestations) | 1 | 0 | 0 | 0
Pyelocystitis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 2 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 1 | 0 | 0
Salmonella sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 10 | 4 | 4 | 8
Septic shock (Infections and infestations) | 5 | 2 | 2 | 3
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 0 | 2 | 0
Tuberculosis (Infections and infestations) | 1 | 3 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1 | 0 | 0
Typhoid fever (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 7 | 6 | 9
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 2 | 3
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral myocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chemical injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 4 | 3
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Exposure via inhalation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 4 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 3
Femur fracture (Injury, poisoning and procedural complications) | 5 | 6 | 5 | 8
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 4 | 1 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint capsule rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 11
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 6 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
VIth nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 1 | 0
Blood glucose fluctuation (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 2 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 2 | 0 | 2
Liver function test abnormal (Investigations) | 0 | 1 | 2 | 0
Myocardial necrosis marker increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 1 | 6 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 6 | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 10 | 11 | 8
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 4 | 3
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 1 | 5
Bladder cancer stage I, without cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 5 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4 | 3
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 1 | 2
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 5 | 4
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Eyelid haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 1
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Gastrointestinal tract adenoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 4 | 4
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 3 | 2
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 3 | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 13 | 17 | 10
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm of choroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 4
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 9 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7 | 0 | 4
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Oesophageal squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 4 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 8 | 11
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 3
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Round cell liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Scrotal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 3 | 6
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 4 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 5 | 12
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vulvar adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Basilar artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 1
Brain mass (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 4 | 6 | 4 | 7
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 3
Cerebellar atrophy (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 3 | 3
Cerebral infarction (Nervous system disorders) | 5 | 6 | 4 | 7
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 16 | 11 | 11 | 18
Cerebrovascular disorder (Nervous system disorders) | 2 | 1 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 2 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Coma (Nervous system disorders) | 0 | 1 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Diplegia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 4 | 4 | 4 | 3
Headache (Nervous system disorders) | 2 | 0 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 2 | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 19 | 15 | 14 | 19
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 1 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Postictal paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 2
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sacral radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 4 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2 | 3 | 1
Syncope (Nervous system disorders) | 6 | 7 | 6 | 10
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 7 | 13 | 16 | 9
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 2
Vascular parkinsonism (Nervous system disorders) | 1 | 0 | 0 | 0
Vertebral artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 1 | 2
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 1 | 2
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 3 | 1 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 7 | 8 | 9
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 4 | 6 | 2 | 4
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 1 | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 4 | 4
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 7 | 2 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 2 | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 4 | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 7 | 3 | 5
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 | 7 | 8 | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 262 | 214 | 245 | 189
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 2 | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 3 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hydrothorax (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3 | 9
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 17 | 13
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9 | 9
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin sensitisation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Finger amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 10 | 8 | 5 | 4
Aortic aneurysm rupture (Vascular disorders) | 1 | 2 | 3 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 1
Aortic disorder (Vascular disorders) | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 1 | 3 | 3
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 3
Arterial rupture (Vascular disorders) | 1 | 0 | 0 | 0
Arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 2
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1 | 2 | 2
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 2 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 6 | 5 | 4 | 5
Diabetic microangiopathy (Vascular disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 3 | 3 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 7 | 9 | 8 | 11
Hypertensive crisis (Vascular disorders) | 3 | 5 | 5 | 9
Hypertensive emergency (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 4 | 8 | 2 | 7
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 2 | 2 | 3 | 2
Intermittent claudication (Vascular disorders) | 1 | 0 | 3 | 0
Leriche syndrome (Vascular disorders) | 0 | 0 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Penetrating atherosclerotic ulcer (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 9 | 16 | 11 | 5
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 4 | 3 | 2 | 0
Peripheral artery thrombosis (Vascular disorders) | 2 | 3 | 1 | 3
Peripheral circulatory failure (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 4 | 3 | 3 | 4
Peripheral vascular disorder (Vascular disorders) | 1 | 8 | 3 | 3
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 0
Renovascular hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Secondary hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0 | 1
Subclavian steal syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 1 | 0 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 2 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
Vascular occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Vascular stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Vessel perforation (Vascular disorders) | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4131) | Fluticasone Furoate 100 µg (N=4157) | Vilanterol 25 µg (N=4140) | Fluticasone Furoate/Vilanterol 100/25 µg (N=4140)
Bronchitis (Infections and infestations) | 165 | 184 | 168 | 166
Influenza (Infections and infestations) | 118 | 116 | 122 | 137
Nasopharyngitis (Infections and infestations) | 310 | 366 | 352 | 367
Upper respiratory tract infection (Infections and infestations) | 194 | 240 | 212 | 262
Back pain (Musculoskeletal and connective tissue disorders) | 140 | 168 | 162 | 173
Headache (Nervous system disorders) | 308 | 332 | 327 | 291
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 969 | 939 | 938 | 779
Cough (Respiratory, thoracic and mediastinal disorders) | 254 | 224 | 215 | 206
Dyspnoea (Nervous system disorders) | 172 | 185 | 132 | 125
Hypertension (Vascular disorders) | 129 | 138 | 124 | 152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.